CLINICAL TRIAL: NCT02148172
Title: Optimizing Plyometric Training for Functional Recovery Post-ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry); American Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Ryan Mizner, Associate Professor, University of Montana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UM IRB 282-13
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Anterior Cruciate Ligament Injury; Knee Injury
Keywords: Knee; plyometrics; motor learning; psychological factors
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Plyometric Training (Active Comparator): Participants will undergo treatment 2 times a week for 8 weeks with plyometric exercises deemed to be consistent with best practice delivered at a standard dosage of sets and repetitions.
  Interventions: Procedure: Standard Plyometric Training
- Plyometric Training with BWS (Experimental): Participants will undergo treatment 2 times a week for 8 weeks with plyometric exercises deemed to be consistent with best practice with a treatment volume of sets and repetitions that exceeds standard practice. Higher number of practice trials will be completed with body weight support (BWS) to reduce load. Participants will start at 30 percent of body weight and will be slowly weaned away over time.
  Interventions: Procedure: Plyometric Training with BWS

INTERVENTIONS:
Procedure: Standard Plyometric Training — Participants will undergo individualized practice exercises of jumping, hopping, and cutting tasks consistent with standard published exercises.
  Arms: Standard Plyometric Training
Procedure: Plyometric Training with BWS — Participants will undergo individualized practice exercises of jumping, hopping, and cutting tasks consistent with standard published exercises while their body weight is supported via adjustable harness.
  Arms: Plyometric Training with BWS

SUMMARY:
While surgical anterior cruciate ligament reconstruction (ACLR) of the knee restores passive stability, studies are showing consistently poor long-term outcomes. Unusually high risks of early-onset osteoarthritis and re-injury, and low rate of return to sport following ACLR all seem to be related to a chronic tendency to land stiff-legged from a jump or hop, which itself may be due to fear of re-injury. Decreased knee bending for force absorption simultaneously decreases performance level and increases risk for injury and arthritic changes.

The purpose of the proposed study is to compare a current best-practice plyometric training program to one utilizing body weight support to increase repetition and improve performance in the initial phases. The investigators hypothesize that we will see larger improvements in absorptive capacity of the knee and better confidence in activity immediately following body weight support training, as well as improved retention of training effects after a two-month period.

ELIGIBILITY:
Inclusion Criteria:

* speak and understand English
* age between 12-35 years
* unilateral anterior cruciate ligament reconstruction between 6-48 months prior
* activity level greater than or equal to level 5 on the Tegner Activity Scale

Exclusion Criteria:

* Weight in excess of 300 pounds (136 kg)
* contralateral/bilateral ACL reconstruction or an unreconstructed ACL injury
* history of a posterior cruciate ligament injury
* lower extremity of back injury or other condition (e.g. cerebral palsy) that has limited their normal activities of daily living within the last 6 months

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in sagittal plane knee kinetics and kinematics | Baseline and after 8 weeks of training
Change in psychological readiness for sports activities via survey scores | baseline and after 8 weeks of training
Change in motor patterning via electromyography of quadriceps and hamstring muscles | Baseline and after 8 weeks of training

SECONDARY OUTCOMES:
Retention of Biomechanical Adaptions in Knee kinetics and kinematics | Change from end of 8 weeks of training to 2 month follow-up
Retention of adaptations in Psychological Readiness for Sport via survey | Change from end of 8 weeks of training to 2 month follow-up
Retention of adaptations in motor patterning via electromyography | Change from end of 8 weeks of training to 2 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ryan L Mizner, PT, PhD, Principal Investigator — University of Montana
Locations (1):
- University of Montana, Movement Science Laboratory, Missoula, Montana, United States

REFERENCES:
- [Derived] Elias ARC, Harris KJ, LaStayo PC, Mizner RL. Clinical Efficacy of Jump Training Augmented With Body Weight Support After ACL Reconstruction: A Randomized Controlled Trial. Am J Sports Med. 2018 Jun;46(7):1650-1660. doi: 10.1177/0363546518759052. Epub 2018 Mar 20. PMID 29558161